CLINICAL TRIAL: NCT01193218
Title: A Double-blind, Randomised, Parallel Group Efficacy and Safety Study of BI 10773 (5 mg, 10 mg, 25 mg, and 50 mg) Compared to Placebo When Administered Orally Once Daily Over 12 Weeks, as Monotherapy, in Patients With Type 2 Diabetes and Insufficient Glycaemic Control Despite Diet and Exercise, Followed by a 40 Week Randomised Extension Study to Assess Long Term Safety of BI 10773 (10 mg and 25 mg)
Brief Title: Empagliflozin (BI 10773) Dose Finder Study in Japanese Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.38
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (5):
- BI 10773 low dose QD (Experimental): BI 10773 tablets low dose once a day
  Interventions: Drug: Placebo (mid dose); Drug: Placebo (high dose); Drug: BI 10773
- BI 10773 mid-low dose QD (Experimental): BI 10773 tablets mid-low dose once a day
  Interventions: Drug: Placebo (high dose); Drug: Placebo (low dose); Drug: BI 10773
- BI 10773 mid-high dose QD (Experimental): BI 10773 tablets mid-high dose once a day
  Interventions: Drug: BI 10773; Drug: Placebo (high dose); Drug: Placebo (low dose); Drug: Placebo (mid dose)
- BI 10773 high dose QD (Experimental): BI 10773 tablets high dose once a day
  Interventions: Drug: Placebo (low dose); Drug: Placebo (mid dose); Drug: BI 10773
- Placebo (Placebo Comparator): Placebo tablets once a day
  Interventions: Drug: Placebo (low dose); Drug: Placebo (high dose); Drug: Placebo (mid dose)

INTERVENTIONS:
Drug: Placebo (low dose) — Placebo tablets once a day
  Arms: Placebo
Drug: Placebo (low dose) — Placebo tablets once a day
  Arms: BI 10773 high dose QD
Drug: Placebo (mid dose) — Placebo tablets once a day
  Arms: BI 10773 low dose QD
Drug: Placebo (high dose) — Placebo tablets once a day
  Arms: BI 10773 low dose QD
Drug: BI 10773 — BI 10773 tablets low dose once a day
  Arms: BI 10773 low dose QD
Drug: Placebo (mid dose) — Placebo tablets once a day
  Arms: BI 10773 high dose QD
Drug: Placebo (high dose) — Placebo tablets once a day
  Arms: Placebo
Drug: Placebo (high dose) — Placebo tablets once a day
  Arms: BI 10773 mid-low dose QD
Drug: BI 10773 — BI 10773 tablets mid-high dose once a day
  Arms: BI 10773 mid-high dose QD
Drug: BI 10773 — BI 10773 tablets high dose once a day
  Arms: BI 10773 high dose QD
Drug: Placebo (mid dose) — Placebo tablets once a day
  Arms: Placebo
Drug: Placebo (high dose) — Placebo tablets once a day
  Arms: BI 10773 mid-high dose QD
Drug: Placebo (low dose) — Placebo tablets once a day
  Arms: BI 10773 mid-low dose QD
Drug: Placebo (low dose) — Placebo tablets once a day
  Arms: BI 10773 mid-high dose QD
Drug: BI 10773 — BI 10773 tablets mid-low dose once a day
  Arms: BI 10773 mid-low dose QD
Drug: Placebo (mid dose) — Placebo tablets once a day
  Arms: BI 10773 mid-high dose QD

SUMMARY:
This study is conducted to determine the most appropriate therapeutic doses of BI 10773 in Japanese patients with T2DM at first treatment period. The second treatment period is required to obtain sufficient safety data (one-year exposure to BI 10773) in Japanese patients with T2DM according to the ICH E1 guideline.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of type 2 diabetes mellitus prior to informed consent
* Male and female patients on diet and exercise regimen who are:

  1. drug-naïve, defined as no antidiabetic drugs for 10 weeks prior to informed consent.
  2. pre-treated with one oral antidiabetic drug; the present antidiabetic therapy has to be unchanged for 10 weeks prior to informed consent.
* HbA1c at Visit 1a:

  1. for patients who are drug naïve: HbA1c >=7.0 to =<10.0%
  2. for patients treated with one oral antidiabetic drug: HbA1c >=6.5 to =<9.0%
* HbA1c of >=7.0% and =<10% at Visit 2 (start of run-in)

Exclusion criteria:

* Uncontrolled hyperglycaemia with a glucose level >240 mg/dL (>13.3 mmol/L) after an overnight fast during wash-out/placebo run-in period and confirmed by a second measurement (not on the same day).
* Acute coronary syndromes, stroke or transient ischaemic attack within 12 weeks prior to informed consent
* Impaired renal function, defined as calculated eGFR <60 ml/min (MDRD formula) during screening and/or wash-out period and/or run-in phase.
* Bariatric surgery within the past 2 years and other gastrointestinal surgeries that induce chronic malabsorption
* Blood dyscrasias or any disorders causing hemolysis or unstable Red Blood Cell (e.g. malaria, babesiosis, haemolytic anemia)
* Treatment with anti-obesity drugs (e.g. sibutramine, mazindol) 12 weeks prior to informed consent or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen, etc.) leading to unstable body weight

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (32):
- Japan (32):
  - 1245.38.016 Boehringer Ingelheim Investigational Site, Chiyoda-ku, Tokyo
  - 1245.38.001 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1245.38.003 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1245.38.002 Boehringer Ingelheim Investigational Site, Hachioji, Tokyo
  - 1245.38.010 Boehringer Ingelheim Investigational Site, Hanamaki, Iwate
  - 1245.38.005 Boehringer Ingelheim Investigational Site, Kamakura, Kanagawa
  - 1245.38.020 Boehringer Ingelheim Investigational Site, Kanazawa, Ishikawa
  - 1245.38.013 Boehringer Ingelheim Investigational Site, Kashiwa, Chiba
  - 1245.38.019 Boehringer Ingelheim Investigational Site, Katsushika-ku, Tokyo
  - 1245.38.021 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 1245.38.024 Boehringer Ingelheim Investigational Site, Matsuyama, Ehime
  - 1245.38.004 Boehringer Ingelheim Investigational Site, Minato-ku, Tokyo
  - 1245.38.011 Boehringer Ingelheim Investigational Site, Moriya, Ibaraki
  - 1245.38.030 Boehringer Ingelheim Investigational Site, Naha, Okinawa
  - 1245.38.032 Boehringer Ingelheim Investigational Site, Okawa, Fukuoka
  - 1245.38.031 Boehringer Ingelheim Investigational Site, Okinawa, Okinawa
  - 1245.38.025 Boehringer Ingelheim Investigational Site, Saga, Saga
  - 1245.38.014 Boehringer Ingelheim Investigational Site, Saitama, Saitama
  - 1245.38.006 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1245.38.007 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1245.38.008 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1245.38.009 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1245.38.012 Boehringer Ingelheim Investigational Site, Sasima-gun, Ibaraki
  - 1245.38.015 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1245.38.018 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1245.38.017 Boehringer Ingelheim Investigational Site, Suginami-ku, Tokyo
  - 1245.38.022 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1245.38.023 Boehringer Ingelheim Investigational Site, Ube, Yamaguchi
  - 1245.38.026 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa
  - 1245.38.027 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa
  - 1245.38.028 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa
  - 1245.38.029 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Shiba T, Ishii S, Okamura T, Mitsuyoshi R, Pfarr E, Koiwai K. Efficacy and safety of empagliflozin in Japanese patients with type 2 diabetes mellitus: A sub-analysis by body mass index and age of pooled data from three clinical trials. Diabetes Res Clin Pract. 2017 Sep;131:169-178. doi: 10.1016/j.diabres.2017.07.004. Epub 2017 Jul 8. PMID 28753486
- [Derived] Kadowaki T, Haneda M, Inagaki N, Terauchi Y, Taniguchi A, Koiwai K, Rattunde H, Woerle HJ, Broedl UC. Efficacy and safety of empagliflozin monotherapy for 52 weeks in Japanese patients with type 2 diabetes: a randomized, double-blind, parallel-group study. Adv Ther. 2015 Apr;32(4):306-18. doi: 10.1007/s12325-015-0198-0. Epub 2015 Apr 7. PMID 25845768

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Empa 10mg: It is actually placebo once daily group in the 12-week first treatment period, and placebo/empagliflozin 10 mg once daily group in the 40-week second treatment period
- Placebo/Empa 25 mg: It is actually N/A in the 12-week first treatment period, and placebo/empagliflozin 25 mg once daily group in the 40-week second treatment period
- Empa 5mg/10mg: It is actually empagliflozin 5 mg once daily group in the 12-week first treatment period, and empagliflozin 5 mg/25 mg once daily group in the 40-week second treatment period
- Empa 5 mg/25 mg: It is actually N/A in the 12-week first treatment period, and empagliflozin 5 mg/25 mg once daily group in the 40-week second treatment period
- Empa 10mg: Empagliflozin 10 mg once daily group both in the 12-week first treatment period and the 40-week second treatment period
- Empa 25mg: Empagliflozin 25 mg once daily group both in the 12-week first treatment period and the 40-week second treatment period
- Empa 50mg\10mg: It is actually empagliflozin 50 mg once daily group in the 12-week first treatment period, and empagliflozin 50 mg/10 mg once daily group in the 40-week second treatment period
- Empa 50 mg/25 mg: It is actually N/A in the 12-week first treatment period, and empagliflozin 50 mg/25 mg once daily group in the 40-week second treatment period
Period: 0-12 Weeks
Arm/Group | Placebo/Empa 10mg | Placebo/Empa 25 mg | Empa 5mg/10mg | Empa 5 mg/25 mg | Empa 10mg | Empa 25mg | Empa 50mg\10mg | Empa 50 mg/25 mg
Started | 109 (It is actually placebo group) | 0 (It is actually N/A) | 110 (It is actually empa 5mg group) | 0 (It is actually N/A) | 109 | 109 | 110 (It is actually empa 50mg group) | 0 (It is actually N/A)
Completed | 100 | 0 | 107 | 0 | 108 | 106 | 107 | 0
Not Completed | 9 | 0 | 3 | 0 | 1 | 3 | 3 | 0
Not completed — Adverse Event | 6 | 0 | 1 | 0 | 0 | 2 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Period: 12-52 Weeks
Arm/Group | Placebo/Empa 10mg | Placebo/Empa 25 mg | Empa 5mg/10mg | Empa 5 mg/25 mg | Empa 10mg | Empa 25mg | Empa 50mg\10mg | Empa 50 mg/25 mg
Started | 50 | 50 | 54 | 53 | 108 | 106 | 54 | 53
Completed | 45 | 50 | 50 | 50 | 104 | 101 | 51 | 49
Not Completed | 5 | 0 | 4 | 3 | 4 | 5 | 3 | 4
Not completed — Adverse Event | 1 | 0 | 1 | 2 | 3 | 3 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 3 | 0 | 0 | 2 | 1 | 2
Not completed — Other reason than above | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo (12 Week): Placebo once daily group in the 12-week first treatment period
- Empa 5mg (12 Week): Empagliflozin 5 mg once daily group in the 12-week first treatment period
- Empa 10mg (12 Week): Empagliflozin 10 mg once daily group in the 12-week first treatment period
- Empa 25mg (12 Week): Empagliflozin 25 mg once daily group in the 12-week first treatment period
- Empa 50mg (12 Week): Empagliflozin 50 mg once daily group in the 12-week first treatment period
- Total: Total of all reporting groups
Arm/Group | Placebo (12 Week) | Empa 5mg (12 Week) | Empa 10mg (12 Week) | Empa 25mg (12 Week) | Empa 50mg (12 Week) | Total
Number analyzed (Participants) | 109 | 110 | 109 | 109 | 110 | 547
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (8.7) | 57.3 (11.2) | 57.9 (9.4) | 57.2 (9.7) | 56.6 (10.3) | 57.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 32 | 25 | 25 | 137
  Male | 80 | 84 | 77 | 84 | 85 | 410

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c After 12 Weeks of Treatment.
Description: The primary endpoint in this study is the change from baseline in HbA1c after 12 weeks of treatment.
Time Frame: baseline and 12 weeks
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo (12 Week) | Empa 5mg (12 Week) | Empa 10mg (12 Week) | Empa 25mg (12 Week) | Empa 50mg (12 Week)
Number analyzed (Participants) | 109 | 110 | 109 | 109 | 110
percentage of HbA1c | 0.30 (0.09) | -0.42 (0.09) | -0.40 (0.09) | -0.65 (0.09) | -0.61 (0.09)
Statistical Analysis 1: Comparison: Placebo (12 Week) vs Empa 5mg (12 Week); Difference calculated as empa 5mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — the analyses were made sequentially compared with placebo from high dose of empagliflozin and the full significant level (5%) was maintained by the hierarchical procedure; 'treatment', 'renal function', and 'number of previous antidiabetic medication' as a fixed effect and baseline HbA1c as a covariate; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-0.87 to -0.57], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Placebo (12 Week) vs Empa 10mg (12 Week); Difference calculated as empa 10mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-0.85 to -0.55], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Placebo (12 Week) vs Empa 25mg (12 Week); Difference calculated as empa 25mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.10 to -0.80], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Placebo (12 Week) vs Empa 50mg (12 Week); Difference calculated as empa 50mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-1.06 to -0.76], Standard Error of Mean 0.08

2. Secondary Outcome: Occurrence of Treat to Target Efficacy Response
Description: Occurrence of treat to target efficacy response, that is an HbA1c of <7.0% after 12 weeks of treatment
Time Frame: baseline and 12 weeks
Population: Full analysis set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (12 Week) | Empa 5mg (12 Week) | Empa 10mg (12 Week) | Empa 25mg (12 Week) | Empa 50mg (12 Week)
Number analyzed (Participants) | 106 | 107 | 105 | 106 | 107
percentage of participants | 2.8 [0.6 to 8.0] | 26.2 [18.1 to 35.6] | 19.0 [12.0 to 27.9] | 32.1 [23.3 to 41.8] | 32.7 [24.0 to 42.5]
Statistical Analysis 1: Comparison: Placebo (12 Week) vs Empa 5mg (12 Week); Odds ratio calculated as the odds of Empa 5mg divided by the odds of placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The model includes 'treatment', 'renal function', 'number of previous antidiabetic medications' and 'continuous baseline HbA1c'; Odds Ratio (OR) = 19.367, 95% CI 2-sided [5.340 to 70.236]
Statistical Analysis 2: Comparison: Placebo (12 Week) vs Empa 10mg (12 Week); Odds ratio calculated as the odds of Empa 10mg divided by the odds of placebo; Test type: Superiority or Other; p = 0.0003, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 10.889, 95% CI 2-sided [2.942 to 40.301]
Statistical Analysis 3: Comparison: Placebo (12 Week) vs Empa 25mg (12 Week); Odds ratio calculated as the odds of Empa 25mg divided by the odds of placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 27.624, 95% CI 2-sided [7.601 to 99.99] — The upper limit of confidence interval is actually >99.99
Statistical Analysis 4: Comparison: Placebo (12 Week) vs Empa 50mg (12 Week); Odds ratio calculated as the odds of Empa 50mg divided by the odds of placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 44.906, 95% CI 2-sided [12.120 to 99.99] — The upper limit of confidence interval is actually >99.99

3. Secondary Outcome: Change From Baseline in FPG
Description: Change from baseline in FPG after 12 weeks of treatment
Time Frame: baseline and 12 weeks
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo (12 Week) | Empa 5mg (12 Week) | Empa 10mg (12 Week) | Empa 25mg (12 Week) | Empa 50mg (12 Week)
Number analyzed (Participants) | 109 | 110 | 109 | 109 | 110
mg/dL | 4.06 (2.88) | -22.65 (2.97) | -25.28 (2.77) | -33.70 (2.92) | -32.54 (2.97)
Statistical Analysis 1: Comparison: Placebo (12 Week) vs Empa 5mg (12 Week); Difference calculated as empa 5mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; treatment, renal function, number of previous antidiabetic medication as fixed effects, baseline fasting plasma glucose, baseline HbA1c as covariates; Mean Difference (Final Values) = -26.70, 95% CI 2-sided [-31.61 to -21.80], Standard Error of Mean 2.50
Statistical Analysis 2: Comparison: Placebo (12 Week) vs Empa 10mg (12 Week); Difference calculated as empa 10mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -29.34, 95% CI 2-sided [-34.25 to -24.42], Standard Error of Mean 2.50
Statistical Analysis 3: Comparison: Placebo (12 Week) vs Empa 25mg (12 Week); Difference calculated as empa 25mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -37.75, 95% CI 2-sided [-42.66 to -32.84], Standard Error of Mean 2.50
Statistical Analysis 4: Comparison: Placebo (12 Week) vs Empa 50mg (12 Week); Difference calculated as empa 50mg minus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -36.60, 95% CI 2-sided [-41.51 to -31.69], Standard Error of Mean 2.50

4. Other Pre Specified Outcome: Confirmed Hypoglycaemic Adverse Events
Description: Number of patients with confirmed hypoglycaemic adverse events
Time Frame: between first drug intake of study medication up to a period of 7 days (inclusive) after the last drug intake of study medication, up to 392 days
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Placebo (12 Week) | Empa 5mg (12 Week) | Empa 10mg (12 Week) | Empa 25mg (12 Week) | Empa 50mg (12 Week)
Number analyzed (Participants) | 109 | 110 | 109 | 109 | 110
participants | 0 | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: between first drug intake of study medication up to a period of 7 days (inclusive) after the last drug intake of study medication, up to 392 days
Groups:
- Empa 10mg (Randomized, 52 Week): Patients randomized to empagliflozin 10mg once daily for 52 weeks
- Empa 25mg (Randomized, 52 Week): Patients randomized to empagliflozin 25 mg once daily for 52 weeks
- Empa 10mg (With at Least One Dose, 52 Week): Patients with at least one dose of empagliflozin 10 mg once daily for 52-week treatment
- Empa 25mg (With at Least One Dose, 52 Week): Patients with at least one dose of empagliflozin 25 mg once daily for 52-week treatment
Arm/Group | Placebo (12 Week) | Empa 5mg (12 Week) | Empa 10mg (12 Week) | Empa 25mg (12 Week) | Empa 50mg (12 Week) | Empa 10mg (Randomized, 52 Week) | Empa 25mg (Randomized, 52 Week) | Empa 10mg (With at Least One Dose, 52 Week) | Empa 25mg (With at Least One Dose, 52 Week)
Serious Adverse Events (participants affected / at risk) | 3/109 | 0/110 | 0/109 | 3/109 | 1/110 | 3/109 | 8/109 | 8/267 | 15/265
Other Adverse Events (participants affected / at risk) | 15/109 | 19/110 | 16/109 | 26/109 | 20/110 | 39/109 | 49/109 | 83/267 | 93/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (12 Week) (N=109) | Empa 5mg (12 Week) (N=110) | Empa 10mg (12 Week) (N=109) | Empa 25mg (12 Week) (N=109) | Empa 50mg (12 Week) (N=110) | Empa 10mg (Randomized, 52 Week) (N=109) | Empa 25mg (Randomized, 52 Week) (N=109) | Empa 10mg (With at Least One Dose, 52 Week) (N=267) | Empa 25mg (With at Least One Dose, 52 Week) (N=265)
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macular hole (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Device dislocation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Carbohydrate antigen 19-9 increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (12 Week) (N=109) | Empa 5mg (12 Week) (N=110) | Empa 10mg (12 Week) (N=109) | Empa 25mg (12 Week) (N=109) | Empa 50mg (12 Week) (N=110) | Empa 10mg (Randomized, 52 Week) (N=109) | Empa 25mg (Randomized, 52 Week) (N=109) | Empa 10mg (With at Least One Dose, 52 Week) (N=267) | Empa 25mg (With at Least One Dose, 52 Week) (N=265)
Nasopharyngitis (Infections and infestations) | 10 | 8 | 9 | 11 | 11 | 30 | 33 | 62 | 63
Pharyngitis (Infections and infestations) | 1 | 0 | 4 | 3 | 2 | 6 | 6 | 11 | 9
Constipation (Gastrointestinal disorders) | 3 | 2 | 0 | 4 | 2 | 1 | 6 | 3 | 10
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 7 | 2 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 0 | 0 | 4 | 4 | 14 | 10
Pollakiuria (Renal and urinary disorders) | 1 | 4 | 1 | 7 | 6 | 1 | 8 | 4 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.